CLINICAL TRIAL: NCT04193280
Title: Does Blood Sugar Level Affect Postoperative Agitations in Outpatient Pediatric Surgery?
Brief Title: Blood Sugar Level and Postoperative Agitations in Pediatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Zeynep Nur Orhon, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: IstanbulMUPediatricAnesthesia
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Delirium
Keywords: Preoperative fasting time,; Blood glucose level; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for blood sugar level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the effect of fasting time and blood glucose levels on postoperative agitations in pediatric patients who will undergo outpatient surgery.

DETAILED DESCRIPTION:
Emergence delirium is a very important clinic phenomenon, characterized by irritability and severe restlessness in children recovering from anesthesia; it may cause injury to the child recovering from anesthesia or to surgical site and may also lead to parents, who witness emergence delirium to question the quality of anesthesia. Postoperative agitaitons, has been noted with the newer, less soluble inhaled agents and emergence delirium has become a serious problem, taken care in postanesthesia care unit for anesthesiologists. Preoperative anxiety, premedication, anesthetic drugs, pain, type of surgery and emergence in a foreign environment are the factors which take part in the development of emergence delirium. Emotional and less social children, the children with anxious parents, children undergoing upper airway surgery are under risk. Detection of children at risk, the use of appropriate adjuvant drugs, strict control of postoperative pain, and accompanying parents to their children in the recovery room are currently the primary measures to prevent recovery agitation. Further studies are required to discover underlying causes and management of emergence delirium.

In this study pre-and postoperative blood glucose values, preoperative fasting times and hemodynamic values of 200 American Society of Anesthesiologists (ASA) physical status I-2 patients will be recorded. At the end of the operation, patients will be evaluated with Modified Aldrete Sedation Scale, FLACC Pain Rating Scale and PAED Agitation Scale. The results obtained will be evaluated with statistical methods and the relationship between preoperative fasting time and blood glucose levels and postoperative agitations will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 2-12 years of age who will undergo outpatient surgery

Exclusion Criteria:

* ASA III-IV patients, patients with congenital malformation and developmental delays, or any neurological or cardiac diseases

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include children between 2-12 years of age who will be operated in the pediatric operating room. Circumcision, inguinal hernia, undescended testis, lymphadenopathy excision, cystoscopy, adenotonsillectomy cases will be included in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood sugar level | 11.1.2019-5.31.2020
  Blood glucose levels will be measured in pediatric patients who will undergo outpatient surgery.
The fasting time | 11.1.2019-5.31.2020
  Fasting time will be recorded.
The change in blood sugar level | 11.1.2019-5.31.2020
  According to the type of operation, the change in blood sugar level will be detected. Correlation of this change with postoperative agitation will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep N Orhon, MD, Principal Investigator — Istanbul Medeniyet University Goztepe Research and Traininig Hospital
Locations (1):
- Istanbul MU Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)